CLINICAL TRIAL: NCT04937907
Title: Efficacy and Safety of Hydroxychloroquine in Patients With X-linked Alport Syndrome in China (CHXLAS)
Brief Title: Study of Hydroxychloroquine in Patients With X-linked Alport Syndrome in China (CHXLAS)
Acronym: CHXLAS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021SPNR001; 2019YLYM06 (Other Grant/Funding Number: Shanghai Children's Hospital)
Record Dates: First submitted 2021-06-17; First posted 2021-06-24 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Alport Syndrome, X-Linked
Keywords: Alport Syndrome; Hydroxychloroquine; Treatment
MeSH Terms: conditions — Nephritis, Hereditary | interventions — Tablets; benazepril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine Cohort (Experimental): Patients in the cohort will receive Hydroxychloroquine(HCQ) throughout the study.Patients administered HCQ by oral at a dose of 6.5mg per kilogram twice a day for 6 months. During treatment with HCQ, patients also received enalapril(5-10mg qd).
  Interventions: Drug: Hydroxychloroquine Sulfate 100 milligram (mg) Tab; Drug: Benazepril hydrochloride 10 milligram (mg) Tab
- Comparator Cohort (Sham Comparator): During treatment with HCQ, Patients randomized to Comparator Cohort only received enalapril(5-10mg qd).
  Interventions: Drug: Benazepril hydrochloride 10 milligram (mg) Tab

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate 100 milligram (mg) Tab — Patients administered HCQ by oral at a dose of 6.5mg per kilogram twice a day at least 6 months.
  Other Names: HCQ
  Arms: Hydroxychloroquine Cohort
Drug: Benazepril hydrochloride 10 milligram (mg) Tab — Patients administered Benazepril by oral at a dose of 5mg or 10mg once a day at least 6 months.
  Other Names: Benazepril

SUMMARY:
This Phase 2 randomized controlled trial will study the safety, tolerability, and efficacy of Hydroxychloroquine in qualified patients with Alport syndrome. The trial will be open-label, randomized, controlled and will enroll up to 50 patients.

DETAILED DESCRIPTION:
This Phase 2 randomized controlled trial will study the safety, tolerability, and efficacy of Hydroxychloroquine in qualified patients with Alport syndrome. The trial will be open-label, randomized, controlled and will enroll up to 50 patients.

Patients in the Phase 2 cohort will be randomized 1:1 to either Hydroxychloroquine Cohort or Comparator Cohort.

All patients in the study will follow the same visit and assessment schedule. Following randomization on Day 1, patients will be scheduled to be assessed during treatment at Weeks 4, 12, and 24. Patients will not receive study drug during a 24-week withdrawal period between Weeks 25 and 48. Patients will also be scheduled to be assessed at an in person follow up visit at Week 36, and 48.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Age 3-18 years old;
* Diagnosis of Alport syndrome by genetic testing (documented mutation in a gene associated with Alport syndrome, including COL4A3, COL4A4, or COL4A5) or histologic assessment using electron microscopy;
* Screening eGFR ≥ 90 mL/min/1.73 m2;
* ACE inhibitor and/or ARB, the dosing regimen should be stable for at least 4 weeks prior to screening;
* No antirheumatic drugs such as hydroxychloroquine have been used;
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures;

Exclusion Criteria:

* Causes of chronic kidney disease aside from Alport syndrome (including but not limited to other heritable disorders leading to chronic kidney disease, diabetic nephropathy, hypertensive nephropathy, lupus nephritis, IgA nephropathy);
* Prior exposure to hydroxychloroquine;
* Ongoing chronic hemodialysis or peritoneal dialysis therapy;
* Renal transplant recipient;
* Any clinically significant illness within 4 weeks before screening or surgical or medical condition (other than Alport syndrome) that could interfere with the subject's study compliance; confound the study results; impact subject safety; or significantly alter the absorption, distribution, metabolism, or excretion of drugs;
* Participation in other interventional clinical studies;
* Known hypersensitivity to any component of the study drug.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in urinary erythrocyte count(/HP) | Baseline to maximum 48 weeks
  To assess the change in urinary erythrocyte count(/HP) from baseline to week 48 for patients receiving active drug, compared to patients in Comparator Cohort.

SECONDARY OUTCOMES:
Change in 24-hour urinary protein quantity | Baseline to maximum 48 weeks
  To assess the change in 24-hour urinary protein quantity from baseline to week 48 for patients receiving active drug, compared to patients in Comparator Cohort.
Change in urinary albumin characterization | Baseline to maximum 48 weeks
  To assess the change in urinary albumin characterization from baseline to week 48 for patients receiving active drug, compared to patients in Comparator Cohort.
Change in urinary albumin to creatinine ratio | Baseline to maximum 48 weeks
  To assess the change in urinary albumin to creatinine ratio from baseline to week 48 for patients receiving active drug, compared to patients in Comparator Cohort.
Change in urinary erythrocyte count(urinary sediment analyzer) | Baseline to maximum 48 weeks
  To assess the change in urinary erythrocyte count(urinary sediment analyzer) from baseline to week 48 for patients receiving active drug, compared to patients in Comparator Cohort.
Change in eGFR from baseline | Baseline to maximum 48 weeks
  To assess the increase in eGFR from baseline to week 48 for patients receiving active drug, compared to patients in Comparator Cohort.
Number of participants with treatment-related adverse events | Baseline to maximum 48 weeks
  Safety will be assessed by monitoring adverse events, physical examinations and clinical laboratory test through 48 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-yan Huang, PhD, Study Director — Shanghai Children's Hospital
Locations (1):
- Shanghai Children's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hertz JM, Thomassen M, Storey H, Flinter F. Clinical utility gene card for: Alport syndrome - update 2014. Eur J Hum Genet. 2015 Sep;23(9). doi: 10.1038/ejhg.2014.254. Epub 2014 Nov 12. No abstract available. PMID 25388007
- [Background] Daga S, Donati F, Capitani K, Croci S, Tita R, Giliberti A, Valentino F, Benetti E, Fallerini C, Niccheri F, Baldassarri M, Mencarelli MA, Frullanti E, Furini S, Conticello SG, Renieri A, Pinto AM. New frontiers to cure Alport syndrome: COL4A3 and COL4A5 gene editing in podocyte-lineage cells. Eur J Hum Genet. 2020 Apr;28(4):480-490. doi: 10.1038/s41431-019-0537-8. Epub 2019 Nov 21. PMID 31754267
- [Background] Schrezenmeier E, Dorner T. Mechanisms of action of hydroxychloroquine and chloroquine: implications for rheumatology. Nat Rev Rheumatol. 2020 Mar;16(3):155-166. doi: 10.1038/s41584-020-0372-x. Epub 2020 Feb 7. PMID 32034323
- [Background] Yang YZ, Chen P, Liu LJ, Cai QQ, Shi SF, Chen YQ, Lv JC, Zhang H. Comparison of the effects of hydroxychloroquine and corticosteroid treatment on proteinuria in IgA nephropathy: a case-control study. BMC Nephrol. 2019 Aug 5;20(1):297. doi: 10.1186/s12882-019-1488-6. PMID 31382914
- [Background] Liu LJ, Yang YZ, Shi SF, Bao YF, Yang C, Zhu SN, Sui GL, Chen YQ, Lv JC, Zhang H. Effects of Hydroxychloroquine on Proteinuria in IgA Nephropathy: A Randomized Controlled Trial. Am J Kidney Dis. 2019 Jul;74(1):15-22. doi: 10.1053/j.ajkd.2019.01.026. Epub 2019 Mar 25. PMID 30922594